CLINICAL TRIAL: NCT03862001
Title: Lung Cancer Screening: A Multilevel Intervention
Acronym: LungCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 17-22564
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Lung Cancer
Keywords: randomized control trial; lung cancer risk assessment; shared decision making
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: The intervention will involve a randomized control trial (RCT) with an intervention group that receives LungCARE and a comparison group that does not receive LungCARE.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LungCARE Group (Experimental): The intervention group will receive the LungCARE intervention
  Interventions: Behavioral: LungCARE
- Comparison Group (No Intervention): The comparison group will receive usual care.

INTERVENTIONS:
Behavioral: LungCARE — The LungCARE intervention involves patient and PCP components. The patient component consists of watching a short, educational video, answering questions about lung cancer screening preferences, and receiving a patient report and handout.
  The PCP component consists of receiving a similar report (physician report) prior to the patient visit. This report is based on the patient's risk factors and lung cancer screening preferences. It contains additional information about documenting discussions related to risk, screening, and referrals in the electronic medical record system.
  Arms: LungCARE Group

SUMMARY:
The study will develop and test the feasibility of the Lung Cancer Assessment of Risk and Education (LungCARE) intervention to increase discussions about lung cancer screening between patients and physicians. This intervention will be designed to reach primary care patients and will be implemented at three levels of the healthcare structure: patient, physician, and system. The patient component includes a short lung cancer screening video and questions regarding screening preferences. Patients will receive immediate feedback in a report (patient report) that summarizes their lung cancer screening preferences and a handout summarizing the educational video. At the physician level, primary care physicians (PCPs) will receive a similar report (physician report), which will be delivered to them prior to the patient visit. The report contains additional information about documenting discussion related to risk, screening, and referrals in the electronic health record (EHR) system (system component). The investigators will develop the LungCARE intervention and have a comparison group that will receive usual care. Preliminary testing of LungCARE will occur via a randomized controlled trial (RCT) at the University of California, San Francisco, General Internal Medicine and Women's Health Primary Care clinics. The RCT will evaluate LungCARE among 50 PCPs and 120 high-risk current and former smoker patients. The investigators will determine whether the intervention is accepted by patients and physicians and whether patients who received LungCARE are more likely to discuss lung cancer screening with their physicians when compared to patients and physicians in the comparison group. The investigators will also determine whether the intervention affects knowledge of lung cancer and low-dose computed tomography (LDCT) screening, perception of risk, and worry about lung cancer in patients when compared to patients in the comparison group. The investigators expect their research to provide specific recommendations that will facilitate patient-physician discussions about LDCT screening and promote shared decision-making among patients and physicians.

ELIGIBILITY:
Inclusion Criteria:

* age 55-80
* smoked at least 30 pack-years in lifetime
* if former smoker, quit smoking within the last 15 years
* English speaker
* no prior history of lung cancer
* did not have a lung cancer screening test within the last year
* PCP does not object to patient's participation
* have a scheduled visit at University of California, San Francisco (UCSF) internal medicine clinics.

Exclusion Criteria:

* speaking a language other than English
* has a history of lung cancer
* had a lung cancer screening test within the last year
* PCP objects to patient's participation.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Discussion of lung cancer risk and LDCT screening with PCP | Over 3 months
  Outcome 1 will be assessed in the follow-up survey, administered within one week following the clinic visit. All patients will answer the following yes/no questions: "During your PCP visit, did you discuss...your personal risk of getting lung cancer/the risks and benefits of screening/how often people should be screened/whether you should be screened?", "Did you discuss smoking cigarettes?", "Did you talk about smoking and the risk of lung cancer?", and "Did your doctor refer you to or order a test for lung cancer screening?" Each question will be looked at individually and summed into a single score (0-7). Higher scores indicate an increased discussion of lung cancer risk and LDCT screening.
  Three months following the clinic visit, the investigators will review the electronic health records for all patients who signed HIPAA forms. Investigators will gather information about discussion of lung cancer risk and documentation, referrals, counseling, and receipt of LDCT screening.
Knowledge of lung cancer screening | Over one week
  Outcome 2 will be assessed in the follow-up survey, administered within one week following the clinic visit. All patients will answer true/false questions addressing various screening topics (e.g. annual lung cancer screening, false negative scans, false positive scans, who should be screened, and radiation exposure). Correct answers will be given a score of 1 and incorrect answers will be given a score of 0. Responses for each question will be added up to a single score, ranging between 0 and 10. Lower scores indicate lower knowledge and higher scores indicate higher knowledge.
Perception of lung cancer risk | Over one week
  Outcome 3 will be measured using an adapted Lerman Cancer Worry Scale. The following question will be asked over the course of one week, both prior to and following the clinic visit: "In your opinion, compared to most people of your same age, sex, and race, what are you chances of getting lung cancer someday?" Participants will use a five-point Likert scale ("much higher" [1], "higher" [2], "about the same" [3], "lower" [4], "much lower" [5]) to answer the questions. A higher score indicates a lower perception of lung cancer risk. Responses will be compared between the baseline and follow-up surveys.

SECONDARY OUTCOMES:
Worry about lung cancer | Over one week
  Outcome 4 will be measured using an adapted Lerman Cancer Worry Scale. The following questions will be asked over the course of one week, both prior to and following the clinic visit: "How worried are you about getting lung cancer someday?", "During the past month, how much has your worry about lung cancer affected your mood?", "During the past month, how much has your worry about lung cancer affected your ability to perform your daily activities?", and "During the past month, how often have you thought about your chances of getting lung cancer?" Patients will use a 5-point Likert scale ("a lot" [1], "somewhat" [2], "a little" [3], "not at all" [4]) to answer the first 3 questions and a 4-point Likert scale ("almost all the time" [1], "often" [2], "sometimes" [3], "not at all or rarely" [4]) to answer the last question. Higher scores indicate a lower perception of risk. Each question will be examined individually. Responses will be compared between the baseline and follow-up surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Celia Kaplan, DrPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Charles C, Gafni A, Whelan T. Shared decision-making in the medical encounter: what does it mean? (or it takes at least two to tango). Soc Sci Med. 1997 Mar;44(5):681-92. doi: 10.1016/s0277-9536(96)00221-3. PMID 9032835
- [Background] Henderson S, DeGroff A, Richards TB, Kish-Doto J, Soloe C, Heminger C, Rohan E. A qualitative analysis of lung cancer screening practices by primary care physicians. J Community Health. 2011 Dec;36(6):949-56. doi: 10.1007/s10900-011-9394-2. PMID 21442338
- [Background] McBride CM, Emmons KM, Lipkus IM. Understanding the potential of teachable moments: the case of smoking cessation. Health Educ Res. 2003 Apr;18(2):156-70. doi: 10.1093/her/18.2.156. PMID 12729175
- [Background] Poghosyan H, Kennedy Sheldon L, Cooley ME. The impact of computed tomography screening for lung cancer on smoking behaviors: a teachable moment? Cancer Nurs. 2012 Nov-Dec;35(6):446-75. doi: 10.1097/NCC.0b013e3182406297. PMID 22209869
- [Background] Bach PB, Mirkin JN, Oliver TK, Azzoli CG, Berry DA, Brawley OW, Byers T, Colditz GA, Gould MK, Jett JR, Sabichi AL, Smith-Bindman R, Wood DE, Qaseem A, Detterbeck FC. Benefits and harms of CT screening for lung cancer: a systematic review. JAMA. 2012 Jun 13;307(22):2418-29. doi: 10.1001/jama.2012.5521. PMID 22610500
- [Background] Stacey D, Legare F, Lewis K, Barry MJ, Bennett CL, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2017 Apr 12;4(4):CD001431. doi: 10.1002/14651858.CD001431.pub5. PMID 28402085
- [Derived] Walsh JME, Karliner L, Smith A, Leykin Y, Gregorich SE, Livaudais-Toman J, Velazquez AI, Lowenstein M, Kaplan CP. LungCARE: Encouraging Shared Decision-Making in Lung Cancer Screening-a Randomized Trial. J Gen Intern Med. 2023 Nov;38(14):3115-3122. doi: 10.1007/s11606-023-08189-1. Epub 2023 Aug 31. PMID 37653203
- See also: U.S. Preventive Services Task Force. USPTF Bulletin: U.S. Preventive Services Task Force Issues Draft Recommendation Statement on Screening for Lung Cancer. U.S. Preventive Services Task Force 2013. — https://www.uspreventiveservicestaskforce.org/Page/Document/RecommendationStatementFinal/lung-cancer-screening
- See also: Center for Medicare and Medicaid Services. Decision memo for screening for lung cancer with low dose computed tomography (LDCT). — https://www.cms.gov/medicare-coverage-database/details/nca-decision-memo.aspx?NCAId=274